CLINICAL TRIAL: NCT05449327
Title: Xarelto for Thromboprophylaxis After Total Hip and Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB2021079
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Venous Thromboembolism; Arthroplasty
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): The participants are provided with Rivaroxaban 10mg
  Interventions: Drug: Rivaroxaban 10 MG
- Control (No Intervention): The participants are provided without antithrombotics

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Patients are randomly divided into two groups. One group receives no prophylaxis with an anticoagulant, the other one receives Rivaroxaban. The dosage of Rivaroxaban is 10 mg given orally once daily starting on the day of the surgery and continuing the following 13 days.
  Other Names: Xarelto
  Arms: Rivaroxaban

SUMMARY:
Venous thromboembolism is a serious complication after total hip replacement (THR) and total knee replacement (TKR). Previous studies have reported the incidence of both asymptomatic and symptomatic deep vein thrombosis (DVT) after TKR were higher in Taiwan than other countries in Asia. Therefore, the usage of prophylactic antithrombotics should be considered. The efficacy and safety of Xarelto (Rivaroxaban) for preventing venous thromboembolism has been proved. However, there is a lack of study using prospective design to evaluate the efficacy and safety of Xarelto after THR and TKR for Taiwanese. In this study, the investigators use a randomized controlled trial design comparing the incidence of DVT, pulmonary embolism, and complications between intervention and control groups.

DETAILED DESCRIPTION:
This parallel study is conducted in a single hospital. The participants are divided into two groups. One group is provided with Xarelto, and the other one group is provided without any prophylactic antithrombotic. To check the presence of a deep vein thrombosis of the lower limb, bilateral sonographic examinations are arranged for all participants preoperatively and at 3 and 14 days postoperatively. One radiologists who was blinded to the nature of the study interpreted the results of the sonographic examination. The present of pulmonary embolism, DVT-related symptoms, and complications are recorded during the 3-months follow-up in orthopedics outpatients. The symptom which associated with DVT is defined as the signs of leg such as unusual pain, edema, swelling, warm skin, and red or discolored skin. Complications related to Xarelto include major bleeding, infection, and non-healing wound. The expected number of participants in each group is 89, which is calculated by G * Power version 3.1. The intention to treat analysis is used in this study. The investigators compare the incidences of DVT, pulmonary embolism, and complications between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Undergo total knee replacement or total hip replacement

Exclusion Criteria:

* Recent antithrombotics use
* A history of a coagulopathy
* Recent thromboembolic disease
* Preoperative deep vein thrombosis screening presents positive
* Age below 20

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Deep vein thrombosis | Up to 3 months after THR and TKR
  The incidence of both asymptomatic and symptomatic deep vein thrombosis
Pulmonary embolism | Up to 3 months after THR and TKR
  The incidence of pulmonary embolism

SECONDARY OUTCOMES:
Complication | Up to 3 months after THR and TKR
  Major bleeding, infection, and non-healing wound

CONTACTS AND LOCATIONS:
Locations (1):
- Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No